CLINICAL TRIAL: NCT06079775
Title: A Phase 1, Open-Label, Drug-drug Interaction, and Randomized, Double-blind, Controlled, Multiple-dose Pharmacokinetics and Safety Study of Xeruborbactam Oral Prodrug (QPX7831) in Combination With Ceftibuten in Healthy Adult Participants
Brief Title: P1, DDI & MAD PK and Safety Study of Xeruborbactam Oral Prodrug in Combo With Ceftibuten in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qpex Biopharma, Inc. (Industry)
Collaborators: Shionogi Inc. (Industry); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Qpex-102
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-06

CONDITIONS: Bacterial Infections
Keywords: beta-lactamase inhibitor
MeSH Terms: conditions — Bacterial Infections | interventions — Ceftibuten

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Controlled, Crossover, ascending single-and multipledose design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: matched oral placebo capsules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Dose Drug-Drug-Interaction Crossover & Multiple Dose Cohorts (Experimental): DDI crossover part of the study, subjects will be enrolled into 3 cohorts of 8 subjects each, Cohorts 1, 2, & 3 respectively.
  All subjects in Cohorts 1, 2, and 3 will receive a single dose of xeruborbactam oral prodrug (XOP) on Day 1. On Day 6, they will receive a single dose of ceftibuten. On Day 9 they will receive a single combined dose of XOP and ceftibuten.
  During the MAD part of the study, subjects will be enrolled into 2 cohorts, Cohorts 4 & 5 respectively.
  Subjects in Cohorts 4 (16 subjects) will receive either a combined dose of XOP and ceftibuten, active ceftibuten, or active XOP.
  Cohort 4 will be dosed BID on Days 1-9, with last dose on the morning of Day 10.
  Subjects in Cohort 5 (15 subjects) will receive active XOP in comb with active ceftibuten which will be admin orally either twice on Day 1 and QD on Days 2-10 (Group 1), BID on Days 1-9 and QD on Day 10 (Group 2), or TID on Days 1-9 and once on Day 10 (Group 3), based on group assignment.
  Interventions: Drug: Xeruborbactam Oral Prodrug; Drug: Ceftibuten
- Placebo Comparator to maintain the blind (Placebo Comparator): During Cohort 4, Xeruborbactam Oral Prodrug Placebo and Ceftibuten placebo will be used to maintain the blind. In Cohort 4, ten (10) subjects in each cohort will receive a combined dose of xeruborbactam oral prodrug and ceftibuten. Three (3) subjects in each cohort will receive active ceftibuten capsules with xeruborbactam oral prodrug placebo capsules. Three (3) subjects in each cohort will receive active xeruborbactam oral prodrug capsules with ceftibuten placebo capsules.
  Interventions: Drug: Xeruborbactam Oral Prodrug Placebo; Drug: Ceftibuten Placebo

INTERVENTIONS:
Drug: Xeruborbactam Oral Prodrug — Experimental
  Other Names: QPX7831
  Arms: Single Dose Drug-Drug-Interaction Crossover & Multiple Dose Cohorts
Drug: Ceftibuten — Experimental
  Arms: Single Dose Drug-Drug-Interaction Crossover & Multiple Dose Cohorts
Drug: Xeruborbactam Oral Prodrug Placebo — Placebo Comparator
  Other Names: QPX7831 Placebo
  Arms: Placebo Comparator to maintain the blind
Drug: Ceftibuten Placebo — Placebo Comparator
  Arms: Placebo Comparator to maintain the blind

SUMMARY:
A Phase 1, Open-Label, Drug-drug Interaction, and Randomized, Double-blind, Controlled, Multiple-dose Pharmacokinetics and Safety Study of Xeruborbactam Oral Prodrug (QPX7831) in Combination with Ceftibuten in Healthy Adult Participants

DETAILED DESCRIPTION:
Qpex Biopharma, Inc. is developing an oral dosage form that delivers Xeruborbactam, a new boron-based beta-lactamase inhibitor with activity against both serine and metallo-beta-lactamases, for oral treatment in combination with a beta-lactam antibiotic.

Ceftibuten is a cephalosporin antibiotic approved in the US for acute exacerbations of chronic bronchitis, acute bacterial otitis media and pharyngitis/tonsillitis.

This Phase 1 study will assess if a PK interaction exists between xeruborbactam oral prodrug and ceftibuten when given in combination at doses of each drug that have previously been shown to be safe. The study will also assess the safety of the combination with dosing over 10 days.

Study Objectives:

1. To assess the safety, tolerability, and PK of single and multiple doses of xeruborbactam oral prodrug and ceftibuten both in combination and alone, in healthy adult participants.
2. To assess whether there is any PK interaction between xeruborbactam oral prodrug and ceftibuten when administered in combination to healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible to be included in the study only if all of the following criteria apply:

Age

1. Participant must be a healthy adult male or female, 18 to 55 years of age (inclusive) at the time of screening.

   Type of Participant and Disease Characteristics
2. Participants who are overtly medically healthy with clinically insignificant screening results (eg, laboratory profiles, medical histories, ECGs, physical examination) as assessed by the investigator, sub-investigator, or medical officer.

   Weight
3. Body mass index (BMI) ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive). Note: BMI = kg/m2 where kg is a weight in kilograms and m2 is a height in meters squared.

   Sex and Contraceptive/Barrier Requirements
4. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   Male participants:

   If male, agree to be sexually abstinent or agree to use 2 approved methods of contraception (refer to inclusion criterion #5) when engaging in sexual activity from study check-in through 30 days following the last administration of the study drug, and to not donate sperm during this same period of time. If the sexual partner is surgically sterile, contraception is not necessary.
5. Female participants:

   Females of childbearing potential must either be sexually abstinent for 14 days prior to Day 1 and agree to remain so through 30 days following the last administration of the study drug, OR have been using (or agree to use) 2 of the following acceptable methods of birth control for the times specified:
   1. Intra-uterine device (IUD) in place for at least 3 months prior to Day 1 through 30 days following the final dosing of the study drug
   2. Barrier method (condom or diaphragm) for at least 14 days prior to Day 1 through 30 days following the final dosing of the study drug
   3. Stable hormonal contraceptive for at least 3 months prior to Day 1 and barrier method (condom or diaphragm) for at least 14 days prior to Day 1 through 30 days following final dosing of the study drug
   4. Surgical sterilization (vasectomy) of partner at least 6 months prior to Day 1

   Informed Consent
6. Capable of giving signed informed consent as described in Appendix 1 Informed Consent Form (Section 10.1.3) that includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Participants will be excluded from the study if any of the following criteria apply:

Medical Conditions

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
2. Documented hypersensitivity reaction or anaphylaxis to any medication, including ceftibuten or other beta-lactam antibiotics (e.g. cephalosporins, penicillins, carbapenems or monobactams) or any excipients used in this formulation.
3. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
4. Females who are pregnant or lactating.
5. Surgery within the past 3 months prior to Day 1 determined by the investigator, sub-investigator, or medical officer to be clinically relevant.
6. Any acute illness within 30 days prior to Day 1.
7. Any other condition or prior therapy, which, in the opinion of the investigator, sub-investigator, or medical officer would make the participant unsuitable for this study.

   Prior/Concomitant Therapy
8. Use of any prescription medication (with the exception of hormonal contraceptives or hormone replacement therapy for females) within 14 days prior to Day 1.
9. Use of any over-the-counter medication, including herbal products, probiotics and vitamins, within the 7 days prior to Day 1. Up to 2 grams per day of paracetamol is allowed for acute events at the discretion of the investigator, sub-investigator, or medical officer.
10. Use of antacids, H2 receptor blockers or proton pump inhibitors 7 days prior to Day 1. This includes calcium carbonate.

    Prior/Concurrent Clinical Study Experience
11. Participation in another investigational clinical trial within 30 days prior to Day 1 or within 5 half-lives of the previous investigational drug, whichever is longer.

    Diagnostic Assessments
12. QTc corrected according to Fridericia's formula (QTcF) interval > 450 msec for males and > 470 for females or history of prolonged QT syndrome at screening or check-in (Day -1).
13. Calculated creatinine clearance < 80 mL/min (Cockcroft-Gault method) at screening or check-in (Day -1).
14. Any clinically significant abnormalities in laboratory values at screening or check-in (Day -1), in particular:

    1. White blood cell count < 3,000/mm3, hemoglobin < 11g/dL
    2. Absolute neutrophil count < 1,200/mm3 or platelet count < 120,000/mm3
    3. Liver function abnormalities at screening or check-in (Day -1) (defined by an elevation in bilirubin, AST, or ALT > ULN for participants based on age and sex)

    Other Exclusion Criteria
15. Blood donation or significant blood loss (ie, > 500 mL) within 56 days prior to Day 1.
16. Plasma donation within 7 days prior to Day 1.
17. Positive urine drug/alcohol testing at screening or check-in (Day -1).
18. History or presence of alcoholism or drug abuse within the 2 years prior to Day 1.
19. Use of more than 5 packs/week of cigarettes (or equivalent amount of nicotine-containing product) within 6 months prior to Day 1. Use of all nicotine containing products 48 hours prior to admission to clinical research unit. Participants must agree to refrain from smoking for the duration of the study.
20. Excessive intake of alcohol, defined as an average daily intake of > 2 standard drinks for women and > 4 standard drinks for men, (standard drink is the equivalent to 4 oz of wine (approximately 12% abv), 12 oz of regular beer (approximately 5% abv), or 1.5 oz of spirits (80 proof).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment -Emergent Adverse events by subject and by cohort (single dose, multiple doses) | 16 days
  Number of patients with Treatment-Emergent Adverse Events by subject, by cohort, severity and relationship to treatment
Number of patients with changes from baseline in safety parameters | 16 days
  Number of patients with changes in safety parameters before and after dosing by subject and cohort
Peak plasma Concentration measurements by subject and by cohort (Cmax) | 16 days
  Comparison will be performed between the cohorts for concentration measurements (Cmax). Mean graphical presentation of the data will be reported.
  Statistical analysis of exposure parameters will be performed.
Time concentration data measurements by subject and by cohort (Tmax) | 16 days
  Comparison will be performed between the cohorts for time concentration data measurements (Tmax)
Area under the plasma concentration versus time curve (AUC) between cohorts | 16 days
  Comparison will be performed between the cohorts for area under the plasma concentration versus time curve (AUC). Mean graphical presentation of the data will be reported.
  Statistical analysis of exposure parameters will be performed.
Urine Pharmacokinetic (PK) amount excreted by subject and by cohort | 16 days
  Urine Pharmacokinetic (PK) parameters such as amount excreted will be calculated from urinary excretion data
Urine Pharmacokinetic (PK) % dose excreted by subject and by cohort | 16 days
  Urine Pharmacokinetic (PK) parameters such as amount of % dose excreted will be calculated from urinary excretion data

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Loutit, MBChB, Study Director — Qpex Biopharma, Inc.
Locations (1):
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No